CLINICAL TRIAL: NCT03479749
Title: Prospective, Randomized, Double-blind, Placebo-controlled Clinical Trial to Assess the Efficacy and Safety of Intra-articular Injection of RegenoGel-OSP and RegenoGel as a Treatment of Osteoarthritis (OA)
Brief Title: The Effect of Intra-Articular Injection of RegenoGel-OSP™ (Self-Plasma) and RegenoGel™ on Knee Pain in People Suffering From Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ProCore Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PROC-2
Record Dates: First submitted 2018-03-12; First posted 2018-03-27 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- RegenoGel-OSP - RegenoGel-OSP (Experimental): First injection- the patients will receive RegenoGel-OSP; Second injection (after 3 months interval)- the patients will receive RegenoGel-OSP also
  Interventions: Device: RegenoGel-OSP, RegenoGel
- RegenoGel - RegenoGel (Experimental): First injection- the patients will receive RegenoGel; Second injection (after 3 months interval)- the patients will receive RegenoGel also
  Interventions: Device: RegenoGel-OSP, RegenoGel
- Placebo - RegenoGel-OSP (Placebo Comparator): First injection- the patients will receive Placebo; Second injection (after 3 months interval)- the patients will receive RegenoGel-OSP
  Interventions: Device: RegenoGel-OSP, RegenoGel
- Placebo - RegenoGel (Placebo Comparator): First injection- the patients will receive Placebo; Second injection (after 3 months interval)- the patients will receive RegenoGel
  Interventions: Device: RegenoGel-OSP, RegenoGel

INTERVENTIONS:
Device: RegenoGel-OSP, RegenoGel — RegenoGel-OSP (A) and RegenoGel (B) are visco-supplements intended for the intra-articular treatment of OA.

SUMMARY:
This study evaluates the efficacy of intra-articular administration of RegenoGel-OSP™ and RegenoGel™ to treat knee pain and effect on subject's activity and quality of life. During the study the subjects will receive two treatments at a 3-month interval. The study is double-blinded. The subjects will be randomized and sequentially assigned to RegenoGel-OSP™, RegenoGel or placebo treatment in the first treatment. In the second treatment after interval of three months all the subjects will necessarily receive one of the two active products. The follow-up period will continue for one year after first treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has signed and dated the informed consent form
2. Subject is a male or female between 55≤ and ≤ 80 years of age
3. Subject is experiencing pain in the intended study knee with an average VAS score of ≥ 5 over the last week prior to screening.
4. Subject with degenerative changes in the intended study knee that can be categorized as grade II-IV Kellgren Lawrence based upon standing posterior-anterior and lateral radiographs of the knee. This grade will be determined by the physician discretion and also by the Computerized, Automated X-ray-based Scoring and determination of Kellgren Lawrence software. Both methods should indicate a KL grade between II-IV in order for a subject to be eligible for the study.
5. Subject has a Body Mass Index (BMI) between 18.5 and 35

Exclusion Criteria:

1. Subjects with history of significant knee trauma to the intended study knee or with previous arthroscopic surgery of the intended study knee within the last 3 months preceding screening.
2. Subject is experiencing pain in both knees with a VAS score of ≥ 5.
3. Subject had any intra-articular injections to the intended study knee within 3 months prior to Screening.
4. Subject has less than 12-month life-expectancy.
5. Subject is on chronic administration of pain medications (especially opioid pain relievers) and is unable to stop them from the day before each study visit through completion of the study visit.
6. Subject has a history of Psoriatic Arthritis, Rheumatoid Arthritis or any other inflammatory condition associated with arthritis
7. Subject has a wound in the area of the intended study knee
8. Subject has fever signs or symptoms of systemic infection or infection of the intended study knee, on the day before or the day of administration of treatment or placebo.
9. Subject has known sensitivity to any of the treatment components, egg, rubber or latex
10. Subject has a history of anaphylactic shock or other severe systemic response or other adverse event to human blood products
11. Subject has known Human Immunodeficiency Virus / Acquired Immunodeficiency Syndrome (HIV/AIDS), Hepatitis B or C viral infections, or acute or chronic liver disease
12. Subject has ever had cellulitis of the lower extremities, a peripheral vascular disease, or a personal history of clotting disorders.
13. Subject has had cancer in the past 3 years or surgery involving the chest, abdomen, pelvis, or lower extremities in the past year
14. Subject received any treatment with investigational device or product within 30 days prior to Visit l
15. Subject has any recent (acute) or chronic medical, psychiatric, or social problem that might: 1) interfere with the Subject's performance or completion of the trial; 2) obfuscate the Subject's study data; or 3) render the Subject unable to understand the nature, scope, and possible consequences of the study
16. Subject is receiving an antiplatelet and/or anticoagulation medicines (other than Aspirin)
17. Subject ever abused drugs or alcohol (self-reported)
18. Subject received a blood transfusion within 6 months prior to Screening.
19. Subject donated blood or blood products within 3 months prior to Screening
20. Subject has any elective surgery of any kind to the lower extremities or elective surgery requiring general anesthesia scheduled during the course of the trial
21. Subject suffering from severe form of grade KL4 such as total cartilage loss with "bone on bone" as determined by the investigator or by the Computerized, Automated X-ray-based Scoring software.
22. Subject suffering from severe OA and is not able to walk due to pain
23. Pregnant or lactating woman

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2018-02-07 (Actual); Primary Completion 2019-03-04 (Actual); Study Completion 2019-03-04 (Actual)

PRIMARY OUTCOMES:
Efficacy assessment on change in pain in the affected knee joint in response to treatment using the Visual Analog Score (VAS) | Three months
  Change in pain in the effected knee joint in response to treatment using the Visual Analog Score (VAS). VAS score is measured according to the patient's pain rating scale from 1 to 10. The scale of pain increases with increasing pain. For example, score 1 indicates absence of pain (minimum score) and score 10 indicates unbearable pain (maximum score). Each VAS score amounts to only one number of outcome from 1 to 10. VAS will be determined in resting position and in active position. No subscales are combined here.
Efficacy assessment on change in pain in the affected knee joint in response to treatment based on the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) score. | Three months
  Change in pain in the affected knee joint in response to treatment based on the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) score (Pain both at rest and during exercise).

SECONDARY OUTCOMES:
Change in pain in the affected knee joint in response to treatment using the Visual Analog Score (VAS) | Six months
  Change in pain in the effected knee joint in response to treatment using the Visual Analog Score (VAS). VAS score is measured according to the patient's pain rating scale from 1 to 10. The scale of pain increases with increasing pain. For example, score 1 indicates absence of pain (minimum score) and score 10 indicates unbearable pain (maximum score). Each VAS score amounts to only one number of outcome from 1 to 10. VAS will be determined in resting position and in active position. No subscales are combined here.
Change in pain in the affected knee joint in response to treatment based on the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) score | Six months
  Change in pain in the affected knee joint in response to treatment based on the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) score (pain both at rest and during exercise).
Change in the subject´s activity in response to treatments based on the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) score | Three and Six months
  Change in the subject´s activity in response to treatments based on the entire Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) score.
Change from baseline in quality of life in response to treatments using the SF-12 health survey. | Three and Six months
  Change from baseline in quality of life in response to treatments using the SF-12 health survey.
Change in Subjective International Knee Documentation Committee score (IKDC). | Three and Six months
  Change in Subjective International Knee Documentation Committee score (IKDC).
Clinical safety and tolerability assessments which will include: incidence, relatedness and severity of treatment-emergent SAE's, UAE's and AE's in the treatment arms. | Up to 12 months post first injection
  Clinical safety and tolerability assessments up to 12 months post 1st injection which will include: incidence, relatedness and severity of treatment-emergent SAE's, UAE's and AE's in the treatment arms.

CONTACTS AND LOCATIONS:
Locations (5):
- Israel (5):
  - Hadassah Medical Center, Jerusalem
  - Shaare Zedek, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Assaf Harofe Medical Center, Zrifin